CLINICAL TRIAL: NCT00992082
Title: Local Infiltration Analgesia or Intrathecal Morphine in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Professor Kjell Axelsson, University Hospital Orebro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAK-Spinal
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Osteoarthritis
Keywords: Postoperative pain; Local Infiltration Analgesia; Knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative | interventions — Ropivacaine; Ketorolac; Epinephrine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group LIA (Active Comparator): Local Infiltration Analgesia
  Interventions: Drug: ropivacaine, ketorolac and epinephrine
- Group M (Active Comparator): Intrathecal morphine
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: ropivacaine, ketorolac and epinephrine — Spinal injection: bupivacaine 17.5 mg (3,5 mL) + 0.25 mL 0.9% saline. Local Infiltration Analgesia: 400 mg ropivacaine, 30 mg ketorolac and 0.5 mg epinephrine (total volume 166 ml) are infiltrated by the surgeon into the soft tissues peri-articularly during the operation. On the first and on the second postoperative morning, 200 mg ropivacaine, 30 mg ketorolac and 0.1 mg epinephrine, total volume 22 ml, are injected intraarticularly via the catheter.
  Arms: Group LIA
Drug: morphine — Spinal injection: bupivacaine 17.5 mg (3.5 mL) + 0.1 mg (0.25 mL) morphine. No intraarticular injections are given.
  Arms: Group M

SUMMARY:
The purpose of this study is to determine whether local infiltration analgesia is more effective than intrathecal morphine in reducing postoperative pain in total knee arthroplasty.

DETAILED DESCRIPTION:
Postoperative pain is often severe following total knee arthroplasty. Spinal anesthesia is a common method in total knee arthroplasty. Adding morphine to the local anesthetic injected intrathecally prolongs the analgetic effect, but may give the usual opioid side effects. The Local Infiltration Analgesia (LIA) technique has proven effective in reducing postoperative pain in total knee arthroplasty. In the LIA technique a long-acting local anesthetic (ropivacaine), a nonsteroidal anti-inflammatory drug (ketorolac), and epinephrine are infiltrated intraoperatively and via an intraarticular catheter postoperatively.

The aim of this study is to evaluate if spinal anesthesia together with the LIA technique provide better postoperative pain relief and mobilization than spinal anesthesia with addition of morphine to the local anesthetic intrathecally. Primary end-point is morphine consumption the first 48 postoperative hours. Secondary end-points are pain intensity, knee function, time to home readiness, hospital stay, side effects and patient satisfaction. Patients are followed up to 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee arthroplasty under spinal anesthesia.
* Aged 40-85 yrs.
* ASA physical status I-III and mobility indicating normal postoperative mobilization.

Exclusion Criteria:

* Known allergy or intolerance to one of the study drugs.
* Serious liver-, heart- or renal decease.
* Rheumatoid arthritis.
* Chronic pain or bleeding disorder.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-05 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | The first 48 postoperative hours

SECONDARY OUTCOMES:
Pain intensity | 0-3 months
Knee function | 0-3 months
Time to home readiness | 0-2 weeks
Hospital stay | 0-2 weeks
Side effects | 0-3 months
Patient satisfaction | 0-3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Orthopedic Surgery, Örebro, Örebro County, Sweden